CLINICAL TRIAL: NCT01756144
Title: rhBMP-2 vs Autologous Bone Grafting for the Treatment of Non-union of the Docking Site in Tibial Bone Transport
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr Jan Vanderstappen, MD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005664-10
Record Dates: First submitted 2012-12-12; First posted 2012-12-25 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Pseudarthrosis
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous bone grafting (Active Comparator): autologous bone of the iliac crest
  Interventions: Device: rhBMP-2
- rhBMP-2 (Experimental): Inductos, recombinant human bone morphogenetic protein
  Interventions: Device: rhBMP-2

INTERVENTIONS:
Device: rhBMP-2

SUMMARY:
When there is a bone defect, bone transport is used to bridge the defect. Frequently, the bone in the docking site (where the transported bone comes together) doesn't heal.

The objective is to study the effectivity of rhBmp-2 (inductos) to stimulate bone healing, in order to find new techniques to treat non-union of long bones.

The method of the study is a randomized controlled trial, to compare rhBMP-2 and autologous bone grafting in stimulating bone healing in the docking site.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with bone transport (Ilizarov technique) and have non-union of the docking site, which is characterized by absence of bridging callus after two months of compression in the docking site.

Exclusion Criteria:

* Allergy for inductos
* active growth,
* malignancy
* infection
* PAD
* pathological fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Bone healing in the docking site | up to 4 months

SECONDARY OUTCOMES:
Infection | up to one year
Edema | up to one year
cancer | up to one year